CLINICAL TRIAL: NCT06857045
Title: A Prospective, Multicenter, Open-label, Randomized Controlled Trial of 3-month Versus 6-month Dual Antiplatelet Therapy After Implantation of NOVA Intracranial Sirolimus-eluting Stent System
Brief Title: Comparison Three vs Six Months of Dual Anti-platelet Therapy After Sirolimus-eluting Stent Implantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Subgroup analysis based on the main study (NCT05692882), not registered separately.
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOVA II-DAPT
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Intracranial Arteriosclerosis; Intracranial Artery Stenosis; Drug-Eluting Stents
Keywords: intracranial drug-eluting stent; symptomatic intracranial artery stenosis (sICAS)
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months DAPT Intervention (Experimental): After implantation of NOVA stents, all subjects in intervention group will be given dual anti-platelet therapy (DAPT) including aspirin and thienopyridines (clopidogrel or ticagrelor) for 3 months.
  Interventions: Device: NOVA intracranial sirolimus-eluting stent system
- 6 months DAPT Intervention (Active Comparator): After implantation of Firehawk coronary stents, all subjects in control group will be given dual anti-platelet therapy (DAPT) including aspirin and thienopyridines (clopidogrel or ticagrelor) for 6 months.
  Interventions: Device: NOVA intracranial sirolimus-eluting stent system

INTERVENTIONS:
Device: NOVA intracranial sirolimus-eluting stent system — The NOVA stent is a sirolimus-eluting stent system designed for intracranial artery stenosis with a rapid exchangeable balloon.

SUMMARY:
This study is a prospective, multicenter, open-label, randomized controlled clinical trial, aims to assess the clinical non-inferiority of 3 months (short-term) vs 6 months (long-term) of Dual Anti-Platelet Therapy (DAPT) in patients after implanted NOVA intracranial sirolimus-eluting stent system. All participants met the inclusion criteria will be 1:1 randomized to 3 months or 12 months of DAPT at index procedure.

DETAILED DESCRIPTION:
This study will recruit 478 subjects with intracranial atherosclerotic stenosis (ICAS) in China. All participants met the inclusion criteria will be 1:1 randomized to 3 months or 6 months of DAPT after implanting NOVA stent. Clinical follow-up will be carried out at 30 days, 3 months, 6 months, 12 months, 1 year, 2 years, 3 years, 4 years and 5 years after index procedure. The primary endpoint is the composite endpoint of any stroke, death and major bleeding (intracranial or systemic bleeding requiring hospitalization, blood transfusion or surgery) at 1 year.

ELIGIBILITY:
Inclusion criteria

1. Males or females between 35 and 80 years of age.
2. Symptomatic intracranial arteriosclerosis stenosis with reference diameter 2.25-4.00mm;.
3. Intracranial artery stenosis (≥70%) conformed by DSA.
4. Subjects who voluntarily participate in the study and sign informed consent form.

Exclusion Criteria:

1. Subjects who have surgery within previous 30 days or plan to perform major surgery in the next 90 days (surgery grade 3 and above).
2. Subjects of acute hemorrhagic stroke within 3 months.
3. Disabling stroke with a baseline mRS score ≥3.
4. Lesion artery with severe calcification and close neighbour stenosis.
5. Non-atherosclerotic diseases (e.g. arterial dissection, Moya Moya disease, vascular inflammatory lesions caused by infection, autoimmune diseases, post-irradiation, postpartum status; developmental or genetic abnormalities such as fibromuscular dysplasia, sickle cell anemia, suspected vasospasm).
6. The ischaemic event that is highly suspected to be due to vascular embolism from an extracranial arterial segment such as ipsilateral neck/chest arterial occlusion) or cardio embolism such as atrial fibrillation, mitral stenosis, left ventricular thrombus, patent foramen ovale, myocardial infarction within 6 weeks, etc.
7. More than 50% stenosis of the supplying artery of the lesion artery: 1) MCA severe stenosis (lesion artery) with more than 50% stenosis of ipsilateral ICA (supplying artery). 2) Basilar artery severe stenosis (lesion artery) with more than 50% stenosis of dominant VA (supplying artery) stenosis.
8. Accompanied by intracranial tumours or intracranial arteriovenous malformations.
9. The patient who is allergy response to heparin, aspirin, clopidogrel, rapamycin, contrast agents, anaesthetics, or drug eluted stent components.
10. Women who are pregnant or lactating.
11. Due to cognitive or emotional disorders or mental illness, the patient who cannot finish the follow-up.
12. Investigators consider the patient who is not suitable for enrolling in the present trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Any stroke, death and major bleeding | 1 year after operation
  Major bleeding was define as intracranial or systemic bleeding requiring hospitalization, blood transfusion or surgery.

SECONDARY OUTCOMES:
Any stroke or death within 30 days or any ischemic stroke from the original culprit intracranial artery beyond 30 days through 12 months after operation. | 1 year after operation
  The primary outcome was a composite of ischemic/hemorrhagic stroke and all-cause death within 30 days, or any ischemic stroke from the original culprit intracranial artery beyond 30 days through 12 months after operation.
Rate of any stroke (hemorrhagic/ischemic stroke) in the target blood supply area or all-cause death at 30 days after operation | 30 days after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke and any death in the target blood supply area.
Rate of any stroke (hemorrhagic/ischemic stroke) in the non-target blood supply area or all-cause death at 30 days after operation | 30 days after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke and any death in the non-target blood supply area.
Rate of TIA at 30 days, 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  Transient ischemic attack (TIA) is a temporary blockage of blood flow to the brain with symptoms last from only a few minutes up to 24 hours.
Rate of any stroke (hemorrhagic/ischemic stroke) in the target blood supply area at 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke in the target blood supply area.
Rate of any stroke (hemorrhagic/ischemic stroke) in the non-target blood supply area at 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke in the non-target blood supply area.
Rate of death (vascular/ non-vascular death) at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The cause of death was classified as vascular or nonvascular and based on information obtained from the family, medical records, and death certificates. Vascular death included death due to stroke, MI, heart failure, pulmonary embolus, cardiac arrhythmia, or other vascular cause.
Rate of symptomatic ISR and Revascularization at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  symptomatic ISR is defined as ISR associated with an ischemic event in the territory. Revascularization is the restoration or improvement of blood supply, and included surgical operation, endovascularization is the restoration or improvement of blood supply, and included surgical operation, endovascular procedures, etc.
Rate of modified Rankin Scale (mRS) at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
EQ-5D score at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after operation
  A health state defined by the descriptive EQ-5D system can be described by a five-digit number, each digit indicating the score of the corresponding dimension. For the description component a subject self-rates their health in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using either a three-level or a five-level scale.
Rate of in-stent restenosis at 1, 2, 3, 4 years and 5 years after operation (Optional) | 1, 2, 3, 4 years and 5 years after operation
  Patients with ≥50% stenosis of the vessel.
Rate of Device defect | within 5 years of whole trial
  Device defects refer to the unreasonable risks that may endanger human health and life safety during the normal use of medical devices in the course of clinical trials, such as label errors, quality problems, failures, etc.
Rate of bleeding events at 1 years after operation | 1 year after operation
  Bleeding was defined according to Bleeding Academic Research Consortium

CONTACTS AND LOCATIONS:
Overall Officials: Lianbo Gao, Principal Investigator — The Fourth Affiliated Hospital of China Medical University; Jianfeng Han, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The Fourth Affiliated Hospital of China Medical University, Ha’erbin, China